CLINICAL TRIAL: NCT00554463
Title: A Phase II Trial of Combined Modality Therapy With Growth Factor Support for Patients With Limited Stage Small Cell Lung Cancer
Brief Title: G-CSF and Pegfilgrastim in Treating Neutropenia in Patients Undergoing Radiation Therapy and Chemotherapy for Limited Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Cancer and Leukemia Group B (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RTOG 0623; CDR0000574000; NCI-2009-00742 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2007-11-06; First posted 2007-11-07 (Estimated); Results first posted 2014-09-29 (Estimated); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Lung Cancer
Keywords: limited stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Filgrastim; pegfilgrastim; Etoposide; Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combined Modality Therapy with Growth Factor Support (Experimental): Concurrent radiation therapy, cisplatin, etoposide, and filgrastim followed by adjuvant cisplatin, etoposide, and pegfilgrastim.
  Interventions: Drug: Filgrastim; Drug: Pegfilgrastim; Drug: Etoposide; Drug: Cisplatin; Radiation: radiation therapy

INTERVENTIONS:
Drug: Filgrastim — 5 mcg/kg/day IV (intravenous) days 4-13 and days 25-34 for a total of 20 doses.
Drug: Pegfilgrastim — 6 mg via subcutaneous injection days 46 and 67
Drug: Etoposide — Concurrent: 120 mg/m^2, IV on days 1-3 and days 22-24. Adjuvant: 120 mg/m^2, IV on days 43-45 and days 65-66.
Drug: Cisplatin — Concurrent: 60 mg/m^2, IV on days 1 and 22. Adjuvant: 60 mg/m^2, IV on days 43 and 64.
Radiation: radiation therapy — A total of 61.2 Gy in 5 weeks: Once-daily 1.8 Gy fractions for 15 fractions over 3 weeks beginning on day 1 of chemotherapy, then twice-daily 1.8 Gy fractions for 10 fractions over 2 weeks.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cisplatin and etoposide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Colony-stimulating factors, such as G-CSF or pegfilgrastim, may increase the number of immune cells found in bone marrow or peripheral blood and may help the immune system recover from the side effects of chemotherapy and radiation therapy.

PURPOSE: This phase II trial is studying G-CSF and pegfilgrastim to see how well they work in treating neutropenia in patients undergoing combination chemotherapy and radiation therapy for limited stage small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the safety and efficacy of filgrastim (G-CSF) in reducing grade 4 neutropenia or grades 3-4 febrile neutropenia in patients with limited stage small cell lung cancer treated with radiotherapy and concurrent chemotherapy comprising cisplatin and etoposide.

Secondary

* To evaluate the safety and efficacy of pegfilgrastim in reducing grade 4 neutropenia or grades 3-4 febrile neutropenia in patients treated with adjuvant chemotherapy comprising cisplatin and etoposide.
* To estimate the incidence of dose modifications or treatment delays in patients treated with this regimen.
* To estimate the incidence of esophagitis, pneumonitis, and other non-hematological adverse events in patients treated with this regimen.
* To estimate the incidence of grade 4 thrombocytopenia in patients treated with this regimen.
* To estimate the median and two-year rate of progression-free and overall survival of patients treated with this regimen.

After completion of study therapy, patients are followed every 3 months for one year, every 6 months for 2-3 years, and then annually for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed small cell carcinoma of the lung

  * Limited stage disease, defined as any of the following:

    * Tumor confined to one hemithorax
    * T4 tumor not based on malignant pleural effusion
    * N3 disease not based on contralateral supraclavicular involvement
* No complete tumor resection
* Measurable or evaluable disease
* Pleural effusion allowed provided the following conditions are present:

  * Effusion is too small to tap under CT guidance and is not evident on chest x-ray
  * Effusion appears only after a thoracotomy or other invasive procedure
* Must have certification by a Radiation Oncologist that the tumor can be encompassed by limited radiotherapy fields without significantly compromising pulmonary function
* No distant metastases

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-1
* ANC (absolute neutrophil count) ≥ 1,800 cells/mm³
* Platelet count ≥ 100,000 cells/mm³
* Hemoglobin ≥ 10.0 g/dL (transfusion or other intervention to achieve hemoglobin ≥ 8.0 g/dL allowed)
* Total bilirubin ≤ 1.5 mg/dL
* AST (aspartate aminotransferase) or ALT (alanine amino transferase ) ≤ 2 times the upper limit of normal (ULN)
* Alkaline phosphatase < 2.5 times ULN (< 5 times ULN if judged by the investigator to be related to liver metastases)
* Serum creatinine ≤ 1.5 mg/dL
* Creatinine clearance ≥ 50 mL/min
* FEV1 (Forced Expiratory Volume) obtained pre- or post-bronchodilator must be ≥ 1.5 liters/second
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 60 days after the last study treatment
* No prior invasive malignancy, except non-melanomatous skin cancer or other micro-invasive malignancy, or carcinoma in situ of the breast, oral cavity, or cervix, unless the patient has been disease-free for a minimum of 3 years
* No weight loss > 5% for any reason within the past 3 months
* No severe, active comorbidity, defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the past 6 months
  * Transmural myocardial infarction within the past 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics
  * Chronic Obstructive Pulmonary Disease exacerbation with FEV1 (forced expiratory volume) < 1.5 liters/second or other respiratory illness requiring hospitalization or precluding study therapy within the past 30 days
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects
  * AIDS (HIV testing not required for entry into this protocol)
* No prior allergic reaction to the study drugs

PRIOR CONCURRENT THERAPY:

* No prior systemic chemotherapy for lung cancer

  * Prior chemotherapy for a different cancer is allowed, provided it was completed ≥ 5 years prior to registration
* No prior radiotherapy to the region of the study cancer that would result in overlap of radiotherapy fields
* No concurrent intensity-modulated radiotherapy
* No concurrent amifostine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rogerio C. Lilenbaum, MD, Principal Investigator — Mount Sinai Comprehensive Cancer Center at Mount Sinai Medical Center; Ritsuko U. Komaki, MD, FACR, Study Chair — M.D. Anderson Cancer Center; Michael A. Samuels, MD, Study Chair — CCOP - Mount Sinai Medical Center; Jeffrey Crawford, MD, Study Chair — Duke Cancer Institute
Locations (14):
- United States (14):
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Cancer Research UK Medical Oncology Unit at Churchill Hospital & Weatherall Institute of Molecular Medicine - Oxford, Salem, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - McGlinn Family Regional Cancer Center at Reading Hospital and Medical Center, Reading, Pennsylvania
  - Veterans Affairs Medical Center - Milwaukee, Milwaukee, Wisconsin

REFERENCES:
- [Background] Lilenbaum R, Samuels M, Taffaro-Neskey M, Cusnir M, Pizzolato J, Blaustein A. Phase II trial of combined modality therapy with myeloid growth factor support in patients with locally advanced non-small cell lung cancer. J Thorac Oncol. 2010 Jun;5(6):837-40. doi: 10.1097/JTO.0b013e3181d6e141. PMID 20421820

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Combined Modality Therapy With Growth Factor Support
Started | 5
Completed (Subjects contributing any data to results are considered to have completed the study) | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All eligible patients.
Arm/Group | Combined Modality Therapy With Growth Factor Support
Number analyzed (Participants) | 5
Age, Continuous [Median (Full Range); unit: years] | 67 [60 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Grade 3-4 Febrile Neutropenia During Concurrent Chemoradiotherapy
Description: Adverse events were graded using the Common Terminology Criteria for Adverse Events (CTCAE) v3.0. Grade refers to the severity of the AE. The CTCAE v3.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild, Grade 2 Moderate, Grade 3 Severe, Grade 4 Life-threatening or disabling, Grade 5 Death related to AE. No testing was done due to early study termination.
Time Frame: From start of treatment to end of concurrent chemoradiation, for a maximum of 45 days
Population: All registered patients
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Modality Therapy With Growth Factor Support
Number analyzed (Participants) | 5
Participants | 0

2. Secondary Outcome: Number of Patients With Grade 3-4 Febrile Neutropenia During Adjuvant Chemoradiotherapy
Description: Adverse events were graded using the Common Terminology Criteria for Adverse Events (CTCAE) v3.0. Grade refers to the severity of the AE. The CTCAE v3.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild, Grade 2 Moderate, Grade 3 Severe, Grade 4 Life-threatening or disabling, Grade 5 Death related to AE.
Time Frame: From the start to the end of adjuvant chemotherapy, a maximum of 24 days
Population: All registered patients
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Modality Therapy With Growth Factor Support
Number analyzed (Participants) | 5
Participants | 1

3. Secondary Outcome: Number of Patients With Dose Modifications or Treatment Delays
Time Frame: From start of treatment to end of treatment, for a maximum of 66 days
Population: All registered patients
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Modality Therapy With Growth Factor Support
Number analyzed (Participants) | 5
Participants | 2

4. Secondary Outcome: Number of Patients With Grade 3+ Esophagitis, Pneumonitis, and Other Non-hematological Adverse Events
Description: as for outcome 1
Time Frame: From registration to last follow-up, a maximum of 32.9 months
Population: All registered patients
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Modality Therapy With Growth Factor Support
Number analyzed (Participants) | 5
Participants
  Grade 3+ Esophagitis | 0
  Grade 3+ Pneumonitis | 1
  Grade 3+ Other non-hematologic | 1

5. Secondary Outcome: Number of Patients With Grade 4 Thrombocytopenia
Description: as for outcome 2
Time Frame: From registration to last follow-up, a maximum of 32.9 months
Population: All registered patients
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Modality Therapy With Growth Factor Support
Number analyzed (Participants) | 5
Participants | 0

6. Secondary Outcome: Overall Survival
Description: Overall survival time is defined as time from registration/randomization to the date of death from any cause. Overall survival rates are estimated by the Kaplan-Meier method. Patients last known to be alive are censored at the date of last contact. Due to early termination with few patients, only counts of events have been calculated.
Time Frame: From registration to last follow-up, a maximum of 32.9 months
Population: All registered patients
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Modality Therapy With Growth Factor Support
Number analyzed (Participants) | 5
Participants | 3

7. Secondary Outcome: Progression-free Survival
Description: Progression is defined as any failure per Response Evaluation Criteria in Solid Tumors (RECIST) 1.0. Progression-free survival time is defined as time from registration to the date of first progression, death, or last known follow-up (censored). Progression-free survival rates are estimated using the Kaplan-Meier method. Due to early termination with few patients, only counts of events have been calculated.
Time Frame: From registration to last follow-up, a maximum of 32.9 months
Population: All registered patients
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Modality Therapy With Growth Factor Support
Number analyzed (Participants) | 5
Participants | 3

ADVERSE EVENTS:
Description: Patients experiencing more than one of a given adverse event are counted only once for that adverse event.
Arm/Group | Combined Modality Therapy With Growth Factor Support
Serious Adverse Events (participants affected / at risk) | 2/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combined Modality Therapy With Growth Factor Support (N=5)
Blood disorder (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Hemoglobin decreased (Blood and lymphatic system disorders) | 1
Fatigue (General disorders) | 1
Sepsis [with Grade 3-4 ANC] (Infections and infestations) | 1
Neutrophil count decreased (Investigations) | 1
Neurological disorder NOS (Nervous system disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Combined Modality Therapy With Growth Factor Support (N=5)
Atrial flutter (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 2
Esophagitis (Gastrointestinal disorders) | 3
Gastrointestinal disorder (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Salivary gland disorder (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 3
Bronchitis [with Grade 3-4 ANC] (Infections and infestations) | 1
Sepsis [with unknown ANC] (Infections and infestations) | 1
Neutrophil count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
This study stopped accrual early due to unmet targeted accrual goals with 5 subjects accrued out of 44 planned

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.